CLINICAL TRIAL: NCT03055182
Title: Oxygenation of Paravertebral Muscles During Exercise in Chronic Low Back Pain Patients
Acronym: OXYLOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2015_58; 2016-A01151-50 (Other: ID_RCB Number)
Record Dates: First submitted 2017-02-07; First posted 2017-02-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Rehabilitation Program; Muscular Weakness
Keywords: Isokinetic; oxygenation; deoxygenation; aerobic metabolism
MeSH Terms: conditions — Low Back Pain; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low back pain patients (Experimental): Subjects included in physical rehabilitation program.
  Interventions: Other: Physical rehabilitation program
- Control subjects (No Intervention): No intervention administered

INTERVENTIONS:
Other: Physical rehabilitation program — Patients participate during 4 weeks to a physical rehabilitation program.
  Arms: Low back pain patients

SUMMARY:
The study evaluate paraspinal aerobic metabolism of chronic low back pain patients and healthy people during an original and standardized isokinetic protocol.

The aim of this study is to determine a potential alteration of muscular aerobic metabolism in low back pain patients, in order to establish the underlying cause of pain and muscular fatigability characterizing low back pain patients. Then, the aim is to determine if functional rehabilitation program can improve it.

the unit of care have access to metabolic adaptations in measuring the muscular oxygenation and the pulmonary oxygen consumption, using near infrared spectroscopy and gas analyser.

ELIGIBILITY:
Inclusion Criteria:

* For Low back pain patients: suffering from low back pain for at least 3 month
* For control subject: no back pain in the past year

Exclusion Criteria:

* Chronic cardiovascular, pulmonary, metabolic, neurologic disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Deoxyhemoglobin | 20 minutes
  Expressed in arbitrary unit, at rest and during the isokinetic exercises (2 exercises of 5 minutes)

SECONDARY OUTCOMES:
Oxygen consumption | 20 minutes
  Measured in mL/min/kg, at rest and during the isokinetic exercises (2 exercises of 5 minutes)
Work rate | 10 minutes
  Total work measured by the dynamometer in Joules during each exercises
Rate of perceived exertion | 10 minutes
  Bases on the Borg's Scale, evaluating the perceived exertion on a scale from 6 to 20
Pain | 10 minutes
  Bases on a visual analogic scale evaluating the pain on a scale from 0 to 10
Muscular blood volume | 20 minutes
  Expressed in arbitrary unit, at rest and during the isokinetic exercises (2 exercises of 5 minutes)
Sorensen test | 20 minutes
  test is a timed measure used to assess the endurance of the trunk extensor muscles. It is used to assist in the prediction of the incidence and occurrence of low back pain in patients.

CONTACTS AND LOCATIONS:
Overall Officials: André Thevenon, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swyngedhauw, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No